CLINICAL TRIAL: NCT01847417
Title: An Open Label, Balanced, Randomized, Three-treatment, Three-period, Six-sequence, Cross-over, Single Dose, Comparative Bioavailability Pilot Study of Two Test Formulations of Fixed Dose Combination Capsules of Acetylsalicylic Acid (ASA) and Pantoprazole (Each Capsule Contains ASA 100 mg and Pantoprazole 20 mg) Manufactured by Piramal Healthcare Limited, India for GSK Comparing With Aspirin® Protect 100 mg Tablets by Bayer Vital GmbH, and Protium® 20 mg Gastro-resistant Tablets by Nycomed GmbH, in Healthy, Adult, Human Subjects, Under Fed Conditions
Brief Title: Comparative Bioavailability Study of Two Test Products of Fixed Dose Combination Capsule of Acetylsalicylic Acid (ASA) and Pantoprazole (Each Capsule Contains ASA 100 mg and Pantoprazole 20 mg) Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Piramal Clinical Research (Hyderabad, India) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 116498
Record Dates: First submitted 2013-05-02; First posted 2013-05-06 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Ulcers, Duodenal and Gastric
Keywords: Acetylsalicylic acid; Pantoprazole; Fixed dose combination
MeSH Terms: conditions — Ulcer | interventions — Pantoprazole; Tablets; Tablets, Enteric-Coated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Overall Study Arm (Experimental): All the subjects in this study will take part in 3 treatment periods with one of the following treatments in each period. Subjects will receive all three treatments (one per period) in a random order in fed condition.
  Test 1= Fixed dose combination (FDC) formulation one of a capsule containing ASA 100 mg and pantoprazole 20 mg. Test 2= FDC formulation two of a capsule containing ASA 100 mg and pantoprazole 20 mg. Reference= ASA 100 mg tablet + pantoprazole 20 mg gastro-resistant tablet
  Interventions: Drug: Test 1= ASA 100 mg and pantoprazole 20 mg capsule formulation one; Drug: Test 2= ASA 100 mg and pantoprazole 20 mg capsule formulation two; Drug: ASA 100 mg tablet; Drug: Pantoprazole 20 mg gastro-resistant tablet

INTERVENTIONS:
Drug: Test 1= ASA 100 mg and pantoprazole 20 mg capsule formulation one — Formulation Test 1 of a fixed dose combination capsule of ASA and pantoprazole (Each capsule contains ASA 100 mg and pantoprazole 20 mg) manufactured by Piramal Healthcare Limited, India for GSK
Drug: Test 2= ASA 100 mg and pantoprazole 20 mg capsule formulation two — Formulation Test 2 of a fixed dose combination capsule of ASA and pantoprazole (Each capsule contains ASA 100 mg and pantoprazole 20 mg) manufactured by Piramal Healthcare Limited, India for GSK
Drug: ASA 100 mg tablet — Aspirin® Protect 100 mg tablets (Each tablet contains ASA 100 mg) manufactured by Bayer vital GmbH, 51368 Leverkusen, Germany
Drug: Pantoprazole 20 mg gastro-resistant tablet — Protium® 20 mg gastro-resistant tablets (Each gastro-resistant tablet contains 20 mg of pantoprazole (as sodium sesquihydrate)) marketing authorisation holder Nycomed GmbH, Byk-Gulden-Straβe 2, D-78467, Konstanz, Germany

SUMMARY:
An open label, balanced, randomized, three-treatment, three-period, six-sequence, cross-over, single dose, comparative bioavailability pilot study under fed conditions. For fed condition, after check-in, subjects will receive a standard dinner consisting (1000 - 1200 calories) after which they will be required to fast overnight (for at least 10 hours). Thereafter they will receive a non-vegetarian high calorie, high-fat breakfast (800-1000 calories) before dosing, and a standard meal (1700 - 1900 calories) for lunch, snacks and dinner.

ELIGIBILITY:
Inclusion criteria:

* Healthy human subjects within the age range of 18 to 45 years (both inclusive)
* Non-smokers since at least six months
* Willingness to provide written informed consent to participate in the study
* Body-mass index (BMI) of >=18.5 kilogram per meter square (kg/m^2) and <=24.9 kg/m^2, with body weight not less than 50 kg
* Absence of significant disease or clinically significant abnormal laboratory values on laboratory evaluations, medical history or physical examination during the screening
* Normal 12-lead ECG or one with abnormality considered to be clinically insignificant
* Normal chest X-ray Posterior Anterior (PA) view
* Comprehension of the nature and purpose of the study and compliance with the requirement of the protocol.
* Willing to consume non-vegetarian, high fat breakfast prior to dosing.
* Female Subject is eligible to participate if she is of non-childbearing potential (surgically sterile or post-menopausal for at least 1 year); or of child bearing potential practicing an acceptable method of birth control while in the study and for 14 days after the end of the study, as judged by the investigator(s), such as condoms, foams, jellies, diaphragm, intrauterine device (IUD), or abstinence)
* Male Subjects willing to use an approved form of birth control (a double barrier method like condom with spermicide or condom with diaphragm) while in the study and for 14 days after the end of the study, and agree not to donate sperm during this period.

Exclusion criteria:

* Personal / family history/ past history of allergy or hypersensitivity to ASA or pantoprazole or related drugs
* Any contraindication to anticoagulant therapy
* History of sensitivity to heparin or heparin-induced thrombocytopenia
* Past history of active gastric or duodenal ulcer or esophagitis
* A history of cholecystectomy or biliary tract disease including increased liver function tests of known or unknown etiology
* Subjects who have been diagnosed with Gilbert's syndrome (Elevated Liver Function Test (LFT)'s Serum Glutamate Oxaloacetate Transaminase/ Serum Glutamate Pyruvate Transaminase (SGOT/SGPT) + Bilirubin (total and direct))
* Past history of anaphylaxis or angioedema
* Any history of myopathy
* Female subject not willing to use acceptable method of contraception from the date of screening until 14 days after the end of the study
* Male subject not willing to use acceptable method of contraception from the date of screening until 14 days after the end of the study
* Any major illness in the past three months or any clinically significant ongoing chronic medical illness e.g.congestive heart failure, hepatitis, pancreatitis etc.
* Presence of any clinically significant abnormal values during screening e.g. significant abnormality of LFT, Renal (kidney) Function Test (RFT) etc.
* Any cardiac, renal or liver impairment, any other organ or system impairment
* History of seizure or psychiatric disorders
* Presence of disease markers of human immuno deficiency virus (HIV) 1 and 2, and hepatitis B and C virus
* History of significant alcohol consumption for more than two years, or consumption of more than three alcoholic drinks per day or consumption of alcohol within 48 hours prior to check-in in each period and during the study [one drink is equal to one unit of alcohol [one glass wine, half pint beer, and one measure (one ounce) of spirit].
* Presence of painful erythema, oedema, or ulceration in the oral cavity
* Consumption of xanthine containing derivatives (coffee, tea, cola drinks, chocolate) within 48 hours before check-in of each period
* Use of any recreational drug or a history of drug addiction
* Participation in any clinical trial within the past 3 months
* Inaccessibility of veins in left and right arm
* Donation of blood [one unit or 330 millilitre (mL)] within 3 months prior to study check-in
* History of use of any prescription drug therapy within four weeks or over-the-counter (OTC) drugs within two weeks prior to study check-in or repeated use of drugs within the last four weeks
* History of unusual diet, for whatever reason, e.g. low sodium diet, for 7 days prior to check-in for all the three periods
* History of consumption of grapefruit-containing food or drinks within 7 days prior to the study check-in for all the three periods
* Recent history of dehydration from diarrhoea, vomiting or any other reason within a period of 7 days prior to the study check-in for all the three periods
* Difficulty in swallowing solids like tablets/capsules
* Systolic blood pressure below 100 millimetres of mercury (mm Hg) and above 138 mm Hg, diastolic blood pressure below 60 mm Hg and above 90 mmHg
* Heart rate below 60 beats/minute and above 100 beats/minute
* Temperature below 96.0 degree Fahrenheit (F) and above 98.6 degree F
* Female volunteers demonstrating a positive test for pregnancy during screening or currently breastfeeding

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2013-05-16 (Actual); Primary Completion 2013-07-01 (Actual); Study Completion 2013-07-01 (Actual)

PRIMARY OUTCOMES:
Composite of pharmacokinetic (PK) parameters | During each period at pre-dose, 0.167, 0.333, 0.5, 0.667, 0.833, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 14, 16 and 24 hrs post dose
  The bioavailability of two test products was compared with the reference products after determining the plasma PK parameters: Cmax (maximum measured plasma concentration), Tmax (time of Cmax), AUC0-t (area under the plasma concentration versus time curve from time zero to the last measurable concentration), AUC0-infinity (AUC from zero to infinity), t1/2 (time required for the plasma drug concentration to decrease by one half), Kel (terminal rate constant) and AUC_% Extrap_Obs (residual area in percentage determined by formula) for ASA and pantoprazole in relevant treatments

SECONDARY OUTCOMES:
Tolerability of combined ASA and pantoprazole in subjects during the study | Up to 16 days
  Tolerability of combined ASA and pantoprazole in subjects during the study assessed by adverse events, laboratory tests, vital signs and ECG

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Hyderabad, India

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 116498 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/116498?search=study&search_terms=116498#rs
- Available data/document: Study Protocol: 116498 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 116498 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 116498 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 116498 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 116498 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 116498 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register